CLINICAL TRIAL: NCT01234129
Title: Results of Phase III Study to Assess if Zoledronic Acid Have Antumor Activity in Multiple Myeloma
Brief Title: Stem Cell Transplant and Zoledronic Acid Improve Outcome in Previously Untreated Patients With Multiple Myeloma
Status: Completed | Type: Observational
Sponsor: Instituto Mexicano del Seguro Social (Other Government)
Responsible Party: Agustin Aviles, Senior Researcher, Mexican Institute of Social Security
Other Study IDs: kitty1; kitty2 (Other: Mexican Institute of Social Security)
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2010-11-04 (Estimated); Status verified 2009-12

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; stem cell transplant; zoledronic acid
MeSH Terms: conditions — Multiple Myeloma | interventions — Zoledronic Acid

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- zoledronic acid or not zoledronic acid: patients with multiple myeloma will be treated with cytoreductive therapy following by zoledronic acid or not.
  Interventions: Drug: zoledronic acid
- zoledronic acid or not zoledronic acid: patients with multiple myeloma will be treated with cytoreductive therapy following by stem cell transplant and did not received zoledronic acid
  Interventions: Drug: zoledronic acid
- zoledronic acid: Patients with multiple treated with cytoreductive therapy following by stem cell transplant will be planned to received zoledronic acid
  Interventions: Drug: zoledronic acid

INTERVENTIONS:
Drug: zoledronic acid — zoledronic acid, 4 mg,standard dose,at monthly interval, by 2 years

SUMMARY:
Assess the impact in outcome of the use of zoledronic acid in multiple myeloma.

DETAILED DESCRIPTION:
Assess if the use of zoledronic acid can improve outcome in patients with multiple myeloma whose are treated with cytoreductive therapy and stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

Diagnosis of multiple myeloma No previous treatment Symptomatic High risk (ISS) or stage III ( Durie-Salmon) No severe comorbidities -

Exclusion Criteria:

Pregnancy HIV + Refuse treatment

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple myeloma previously untreated
Sampling Method: Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2002-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
progression-free disease and overall toxicity in myeloma multiple | 3 years
  In patients treated with cytoreductive therapy following by stem cell transplant and that received zoledronic acid by 2 years,they were evaluable for assess antitumor effect of zoledronic acid

SECONDARY OUTCOMES:
skeletal event | 3 years
  evaluate the number of skeletal events in patients with multiple myeloma that received zoledronic acid

CONTACTS AND LOCATIONS:
Overall Officials: Agustin Aviles, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Tertiary reference oncology center, Mexico City, Mexico City, Mexico